CLINICAL TRIAL: NCT03542084
Title: Impact of Endocrinology Auto-triggered E-consults on Glycemic Control
Brief Title: Endocrinology Auto-Triggered e-Consults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel M Horn, Director of Population Health and Quality Improvement, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000683
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Unsolicited e-consult (Experimental): The PCP of intervention arm patients will receive an unsolicited e-consult by an endocrinologist offering clinical guidance on how to optimize the patients' glycemic control
  Interventions: Other: Unsolicited endocrine e-consult
- Control (No Intervention): Control arm patients will receive usual care

INTERVENTIONS:
Other: Unsolicited endocrine e-consult — The PCP for intervention arm patients will receive an unsolicited e-consult from an endocrinologist with recommendations on how to improve glycemic control in the intervention patient
  Arms: Intervention: Unsolicited e-consult

SUMMARY:
Diabetes currently affects 25.8 million people in the U.S. Patients with diabetes are generally managed, at least initially, by a primary care practitioner (PCP). As the prevalence of diabetes continues to rise, PCPs are under increased pressure to achieve recommended glycemic targets. Failure to achieve these targets has been shown to increase clinical complications and cost of care.

Endocrinology referral is common for those patients not meeting A1c goals. Unfortunately, access to specialty endocrinology care is limited and patients routinely wait weeks or months before being seen. Electronic consultation (e-consult) is a new and innovative delivery model that has the potential to provide greater access to specialty care. The current system at Massachusetts General Hospital (MGH) allows PCPs to electively place an e-consult to solicit specialist input. Specialists in turn review the patients chart, relevant data and the clinical question and respond within the electronic medical record. E-consults have been well received by both patients and physicians, not only at MGH, but also across many centers in the US. With that said, the e-consult system remains in its infancy and current literature largely focuses on process metrics without hard clinical end-points.

One way to optimize care for patients with diabetes is to automatically trigger an endocrinology e-consult for those not meeting A1c targets. The goal of this project will be to conduct a rigorous scientific evaluation of auto-triggered e-consults across Massachusetts General Hospitals affiliated primary care practices. The e-consults will be unsolicited and triggered based on inclusion criteria that include a1c and date of last PCP visit. This project will leverage an existing diabetes population health registry that is being used currently for ongoing diabetes care initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with a PCP at Massachusetts General Hospital and HbA1c between 8-10 who have seen their PCP in the office within 18 months

Exclusion Criteria:

* Terminal Illness
* Prior visit with MGH diabetes center
* Prior diabetes e-consult completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 6, 12, and 18 months
  Mean change in HbA1c levels in the patient population

SECONDARY OUTCOMES:
Adoption of e-consult recommendations | 6, 12, and 18 months
  Process measures of adoption of the recommendations provided by the e-consultant
A1c testing frequency | 6,12, and 18 months
  number of patients who receive q6 month HbA1c testing in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Horn, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oseran AS, Rao K, Chang Y, He W, Sikora CE, Wexler DJ, Horn DM. HbA1c-Triggered Endocrinology Electronic Consultation for Type 2 Diabetes Management. J Gen Intern Med. 2022 Apr;37(5):1081-1087. doi: 10.1007/s11606-021-07157-x. Epub 2021 Oct 4. PMID 34608564